CLINICAL TRIAL: NCT05329155
Title: Effectiveness and Safety of Early Administration of Heparin At First Medical Contact for STEMI Patients Undergoing Primary Percutaneous Coronary Intervention: a Multicenter, Prospective, Randomized, Controlled Study
Brief Title: Early Administration of Heparin At FMC for PPCI of STEMI Patients
Acronym: HELP-PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Xiangyang Central Hospital (Other); The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture (Other); Wuhan Central Hospital (Other); People's Hospital of Jingshan (Unknown); Chibi General Hospital (Unknown); Xianning Central Hospital (Other); Hubei University of Medicine (Other); Yichang Central People's Hospital (Other); People's Hospital of Tongcheng (Unknown); Ezhou Central Hospital (Unknown); Xiantao First People's Hospital (Unknown); Songzi People's Hospital (Unknown); Anlu People's Hospital (Unknown); Caidian People's Hospital (Unknown); Jiangxia First People's Hospital (Unknown); Jingzhou Central Hospital (Other); Hubei Zhongshan Hospital (Unknown); Guoyao Dongfeng General Hospital (Unknown); Wuhan Puren Hospital (Other); Shiyan People's Hospital (Unknown); General Hospital of Yangtze River shipping (Unknown); Fifth Hospital in Wuhan (Unknown); CR & WISCO General Hospital (Unknown); Xishui People's Hospital (Unknown); Jiangling People's Hospital (Unknown); Wuhan Third Hospital (Other); Laohekou First Hospital (Unknown); The Central Hospital of Huanggang (Other); Wuhan No.1 Hospital (Other); Hanyang University (Other); Wuxue First People's Hospital (Unknown); Tianmen First People's Hospital (Unknown); Xianning First People's Hospital (Unknown); Wuhan No.6 Hospital (Unknown); Wuhan Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chen Jing, MD, PhD, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WDRY2022-K089
Record Dates: First submitted 2022-03-29; First posted 2022-04-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: STEMI; Primary PCI
Keywords: Heparin; Primary Percutaneous Coronary Intervention; ST-Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Heparin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Administration of Heparin in ER (Experimental): Administration of Heparin (100U/Kg body weight) with loading dose of DAPT (Aspirin 300mg and Ticagrelor 180mg) at first medical contact for STEMI patients intended to perform PPCI.
  Interventions: Drug: Heparin Sodium Injection
- Administration of Heparin in Cathlab (Active Comparator): Administration of Heparin (100U/Kg body weight) in Cathlab after insertion of artery sheath catheter.
  Interventions: Drug: Heparin Sodium Injection

INTERVENTIONS:
Drug: Heparin Sodium Injection — Heparin Sodium Injection (100U/Kg body weight)

SUMMARY:
Heparin is the first choice of anticoagulation drug for primary PCI of STEMI patients. However, the priority of use of hepairn in first medical contact or in Cathlab has not yet studied. Previous study revealed early use of antithrombotic drugs could improve patient's survival. Here we supposed that use of heparin at first medical contact could increase the TIMI flow 3 grade ratio in STEMI patients and improve patient's survival and/or reduce MACE rather than in Cathlab.

DETAILED DESCRIPTION:
This study will recruit 944 STEMI patients undergoing primary PCI with the symptom onset within 12 hours in 36 hospitals in Hubei Province, China. The patients will be 1:1 randomly assigned to the intervention group (IG) and control group (CG). Patients in IG will be intravenously administrated with sodium heparin (100U/Kg) at first medical contact, while patients in CG will be administrated with sodium heparin (100U/Kg) through catheter sheath in the CathLab.

Inclusion Criteria:

STEMI patient; Symptom onset in 12 hours; Intended to perform PPCI. Exclusion Criteria:Active bleeding; Life expectancy less than 1 year; History of heparin-induced thrombocytopenia; Mechanical complication of MI (VSR, acute MR); History of CABG; On Coagulation drugs; CPR before randomization; Pregnant or lactating woman;Refused to sign the Informed Consent Form.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patient; Symptom onset in 12 hours; Intended to perform PPCI

Exclusion Criteria:

* Active bleeding; Life expectancy less than 1 year; History of heparin-induced thrombocytopenia; Mechanical complication of MI (VSR, acute MR); History of CABG; On Coagulation drugs; CPR before randomization; Pregnant or lactating woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1145 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
The TIMI 3 flow of the infarct related artery before PPCI | Coronary angiography, before PPCI，anticipated within 2 hours after randomization
  The TIMI 3 flow of the infarct related artery at diagnostic angiography before PPCI

SECONDARY OUTCOMES:
Major adverse cardiovascular or cerebrovascular event | 30 day and 1 year after randomization
  death, cardiac death, admission for heart failure, myocardial infarction, stent thrombosis, unplanned revascularization, and stroke
Major bleeding | 30 day after randomization
  BARC ≥2
Complete epicardial and myocardial reperfusion after PPCI | within 90min after PPCI
  Thrombolysis in myocardial infarction (TIMI) flow grade (TFG) 3 for epicardial reperfusion and TIMI myocardial perfusion (TMPG) grade 3 for myocardial reperfusion and complete (≥70%) ST-segment resolution of the initial sum of ST-segment elevation (STR) 90 minutes after PPCI.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, PhD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan university, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No